CLINICAL TRIAL: NCT02623504
Title: A Double Blind Study To Evaluate the Dose Tolerance and Safety of Equetro (Carbamazepine) Versus Placebo Followed by a Long-Term Maintenance in Children and Adolescents Aged 10-17 Years With Acute Manic or Mixed Bipolar I Disorder
Brief Title: DB/Maintenance of Equetro (Carbamazepine) in Children With Acute Manic or Mixed Bipolar 1 Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No apparent therapeutic effects that was superior to placebo
Sponsor: Validus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAL-EQP-001
Record Dates: First submitted 2015-11-24; First posted 2015-12-07 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Bipolar Disorder
Keywords: Carbamazepine; Equetro; Bipolar I Disorder; Bipolar I Disorder in Children
MeSH Terms: conditions — Bipolar Disorder | interventions — Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Equetro (Experimental): 200-1200 mg of Equetro (carbamazepine) by mouth given in divided doses in the morning and in the evening. Dosage is titrated in 200 mg increments weekly as needed according to subject response.
  Interventions: Drug: Carbamazepine
- Placebo (Placebo Comparator): Placebo dosage to match the active Equetro treatment given in 2 daily doses in the morning and in the evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carbamazepine — 200-1200 mg by mouth daily given in divided doses in the morning and the evening. Doses are titrated weekly in 200 mg increments based upon subject's response.
  Other Names: Equetro
  Arms: Equetro
Drug: Placebo — Dosage to match active treatment by mouth twice daily in the morning and in the evening.
  Arms: Placebo

SUMMARY:
A phase 4 unequal randomization, double blind study to evaluate the dose tolerance and safety of extended release Equetro (carbamazepine) versus placebo followed by an Open label and long term maintenance treatment in children and adolescents aged 10-17 years diagnosed with acute manic or mixed Bipolar I Disorder

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate under double blind conditions the dose tolerance and safety of extended release Equetro (carbamazepine) versus placebo followed by an open label and long term maintenance treatment on extended release Equetro in children and adolescents aged 10-17 year diagnosed with acute manic or mixed bipolar I disorder. The safety evaluations will be based on the occurrence of treatment-emergent adverse events, laboratory values, physical examination, vital signs ECG and trough serum level of study medication. The secondary objective is to evaluate under double blind conditions the efficacy of extended release Equetro versus placebo followed by an open label and long term maintenance treatment on extended release Equetro in children and Adolescents Aged 10-17 years diagnosed with acute manic or mixed Bipolar I disorder. Efficacy evaluations will be based on the measures of YMRS, CGI-S, CGI-I, CDRS-R. Manic episodes over double blind and open label periods will comprise the use of study medication and duration of night time sleep as monitored using a daily diary. Subject's will be enrolled in the double blind period for two months and evaluated on a weekly basis. Once completing the db phase they will continue on Equetro for long term maintenance for an additional six months. Placebo subject will have the opportunity to continue for another eight months in the study. The first two months will be the titration period as was done in the db phase and then they will have the option to continue in the study for an open long term maintenance for and additional 6 months. During the maintenance period subjects will be evaluated for safety and efficacy on a monthly basis. At the end of the study there will be a 30 day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed and dated informed consent from subject, parents or legal guardians.
* Subject must be willing to participate for the duration of the study (8-10 months)
* Subject must meet DSM-V criteria for a primary diagnosis of bipolar I disorder.
* MINI KID administered and ruled out other psychiatric diagnosis.
* ADHD Rating Scale-IV is ruled negative.
* YMRS Score 20 or greater
* CGI-S score of 4 or greater
* CGI-I Global Evaluation score of 4 or less
* Must be aged between 10 and 17 years
* Male and non-pregnant, non-lactating females who agree to comply with contraceptive requirements
* Functioning at an age appropriate level intellectually as deemed by the Investigator
* Subject has no co-morbid conditions that would affect efficacy, safety or tolerability or in any way interfere with the subject's participation in the study
* Subject, parents and legal guardians are able to and willing to comply with study procedures and restrictions
* Must have a satisfactory medical assessment with no clinically significant abnormalities
* Able to avoid grapefruit and grapefruit juice for the duration of the study

Exclusion Criteria:

* Subject has a current controlled or uncontrolled co-morbid psychiatric that could interfere with clinical assessments or study conduct.
* Naive subjects whose symptoms are being controlled on their prescribed medication(s) will not be eligible to participate.
* History of lack of therapeutic response to an adequate trial of carbamazepine to treat bipolar I disorder
* Believed by the Investigator to be acutely at risk for suicidal or violent behavior towards him/her or others, or a history of a suicide attempt requiring general medical intervention
* Subject's bipolar diagnosis is believed secondary to traumatic injury or another general medical condition.
* A history or known presence of clinically significant cardiovascular, hepatic, hematological, immunological (including human immunodeficiency virus, gastro-intestinal or renal disease or any other unstable medical illness that could affect the action, absorption or disposition of the investigational product, or clinical or laboratory assessments
* A history of aplastic anemia, agranulocytosis or bone marrow depression
* A history of seizure disorder, other than a single childhood febrile seizure\
* A history of severe, unstable asthma
* Currently hospitalized for the treatment of psychiatric symptoms.
* Presence of any mental disorder due to a general medical condition
* Presence of abnormal thyroid function that is not adequately treated in the opinion of the Investigator
* Use of ECT, any investigational drug, CYP450 3A4 inhibitors, antidepressants, anxiolytics, sedative hypnotics, antipsychotics, mood stabilizers, ADHD medications, or clozapine in a specified time period prior to the initiation of the study
* Use of any nutraceutical to include, but not limited to any over the counter herbal preparations e.g. Gingko Biloba, St John's Wort, Kava Kava and Ephedra.
* Positive urine drug screen
* History of alcohol or other substance abuse or dependence as defined by DSM-V (except caffeine or nicotine) within the last 6months
* Female subjects with a positive pregnancy test or who are pregnant, lactating, who are less than 6 months post partum, or who cannot be relied upon to use adequate birth control
* Subjects who have previously been enrolled in the Phase IV Multi-Center , Open-Label Safety and Effectiveness Study of Extended-Release Carbamazepine in the Treatment of Acute Manic or Mixed Bipolar I Disorder and subsequently withdrawn
* Subjects with a body weight of ≤65kg
* Family of investigational site staff

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Dose tolerance and safety of Equetro based on occurrence of adverse events, lab values, physical exams, vital signs, ECG's, and trough serum levels of study medications | Duration of the study (8-10 months)

SECONDARY OUTCOMES:
Efficacy of Equetro in the treatment of children and adolescents aged 10-17 years with acute manic or mixed bipolar I disorder measured using the Young Mania Rating Score (YMRS) | Weekly during the double blind period (8 weeks), monthly during the maintenance period (6-8 months)
Efficacy of Equetro in the treatment of children and adolescents aged 10-17 years with acute manic or mixed bipolar I disorder measured using Clinical Global Impressions - Improvement and Severity (CGI-I, CGI-S) | Weekly during the double blind period (8 weeks), monthly during the maintenance period (6-8 months)
Efficacy of Equetro in the treatment of children and adolescents aged 10-17 years with acute manic or mixed bipolar I disorder measured using the Children's Depression Rating Scale - Revised (CDRS-R) | Weekly during the double blind period, monthly during the maintenance period
Efficacy of Equetro in the treatment of children and adolescents aged 10-17 years with acute manic or mixed bipolar I disorder measured by assessing the subject's manic episodes throughout the study period | Duration of the study (8-10 months)
Efficacy of Equetro in the treatment of children and adolescents aged 10-17 years with acute manic or mixed bipolar I disorder measured by assessing the subject's weekly use of study medication | Weekly for the duration of the study (8-10 months)
Efficacy of Equetro in the treatment of children and adolescents aged 10-17 years with acute manic or mixed bipolar I disorder measured by assessing the duration of subject's nighttime sleep monitored using a diary or e-diary | Weekly for the duration of the study (8-10 months)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Findling, MD, Study Director — John Hopkins - Kennedy Krieger Research; Lawrence Ginsberg, MD, Principal Investigator — Red Oak Psychiatry; Morteza Nadjafi, MD, Principal Investigator — APG Research; Mohd Azfar Malik, MD, Principal Investigator — Psych Care Consultants Research
Locations (4):
- United States (4):
  - APG Research, LLC, Orlando, Florida
  - Kennedy Krieger Institute, Baltimore, Maryland
  - PsychCare Consultants, St Louis, Missouri
  - Red Oak Psychiatry Associates, PA, Houston, Texas